CLINICAL TRIAL: NCT04401722
Title: Clinical Impact of Altitude Level on Surgical Outcomes of Pancreaticoduodenectomy for Periampullary Tumour (Multicenter Study)
Brief Title: Clinical Impact of Altitude Level on Surgical Outcomes of Pancreaticoduodenectomy
Acronym: PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ayman El Nakeeb, gastrointestinal surgical center, Mansoura University, Mansoura University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PD in high altitude
Record Dates: First submitted 2020-05-21; First posted 2020-05-26 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Periampullary Cancer
Keywords: pancreaticodudenctomy; POPF; HIGH ALTITUDE
MeSH Terms: conditions — Altitude Sickness

STUDY DESIGN:
Intervention Model Description: it is a multicenter study Aseer centeral hospital, saudia and from Egypt two centers mansoura university and el menia university The patients distributed into two groups group I (G1) PD underwent in the area at the level of the sea, normal altitude region, and group II (G2) PD underwent in high altitude region.
Who Masked: Outcomes Assessor
Masking Description: OUTCOME ASESSOR
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PD in normal altitude (Active Comparator): PD underwent in the area at the level of the sea, normal altitude region
  Interventions: Procedure: PANCREATICODUDENECTOMY
- PD in high altitude region. (Active Comparator): PD underwent in high altitude region.
  Interventions: Procedure: PANCREATICODUDENECTOMY

INTERVENTIONS:
Procedure: PANCREATICODUDENECTOMY — dissection and removal of periampulary tumour with 3 reconstruction PJ, HJ, and GJ
  Other Names: Whippl,s operation

SUMMARY:
Very few papers examine the effect of living at high altitudes on surgical results of major operations. This research is designed to determine the surgical outcomes of PD for periampullary tumour in high altitudes and normal altitudes.

DETAILED DESCRIPTION:
Many recent studies have suggested multiple risk factors affecting postoperative surgical outcomes of PD; THE research is designed to determine the surgical outcomes of PD for periampullary tumour in high altitudes and normal altitude.

it is a multicenter study Aseer central hospital, Saudia and from Egypt two centers Mansoura university and el Menia university

ELIGIBILITY:
Inclusion Criteria:

* periampulary tumour

Exclusion Criteria:

* liver cirrhosis,
* PG,
* advanced tumour,
* vascular resection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-25 (Actual)

PRIMARY OUTCOMES:
the overall postoperative complications | 30 DAYS
  the overall postoperative complications

SECONDARY OUTCOMES:
blood loss | INTRAOPERATIVE
  blood loss
Pulmonary embolism (PE) | 30 days
  Pulmonary embolism (PE)
hospital mortality | 30 days
  death within 30 days of operation

CONTACTS AND LOCATIONS:
Overall Officials: Ayman E Nakeeb, MD, Principal Investigator — Mansoura University, Gastrointestinal Surgery Center
Locations (1):
- Mahmoud Abd El Wahab, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Yes
it will be available for other researchers
Supporting Information: Study Protocol
Time Frame: 6 month
Access Criteria: elnakeebayman@yahoo.com
URL: http://www.mans.edu.eg/en/

REFERENCES:
- [Background] Dutta V, Singh R, Kumar S, Aggarwal N, Hari Kumar KVS. Profile of pulmonary embolism in service personnel posted at high altitude area. Indian Heart J. 2018 May-Jun;70(3):427-429. doi: 10.1016/j.ihj.2017.08.002. Epub 2017 Aug 18. PMID 29961462
- [Result] El Nakeeb A, Attia M, El Sorogy M, Ezzat H, Shehta A, Salem A, El Gawad MA, Hamed H, Allah TA, El-Geidi AA, Fathy O, El Hefnawy E, Zaghloul A. Laparoscopic Pancreaticodudenectomy for Periampullary Tumor: Should it be a Routine? A Propensity Score-matched Study. Surg Laparosc Endosc Percutan Tech. 2020 Feb;30(1):7-13. doi: 10.1097/SLE.0000000000000715. PMID 31461084
- [Result] El Nakeeb A, El Sorogy M, Hamed H, Said R, Elrefai M, Ezzat H, Askar W, Elsabbagh AM. Biliary leakage following pancreaticoduodenectomy: Prevalence, risk factors and management. Hepatobiliary Pancreat Dis Int. 2019 Feb;18(1):67-72. doi: 10.1016/j.hbpd.2018.10.005. Epub 2018 Oct 28. PMID 30413347
- [Result] Prabhakar A, Chatterjee T, Bajaj N, Tyagi T, Sahu A, Gupta N, Kumari B, Nair V, Kumar B, Ashraf MZ. Venous thrombosis at altitude presents with distinct biochemical profiles: a comparative study from the Himalayas to the plains. Blood Adv. 2019 Nov 26;3(22):3713-3723. doi: 10.1182/bloodadvances.2018024554. PMID 31765479
- See also: Mansoura university — http://www.mans.edu.eg/en/
- Available data/document: Study Protocol: Ayman El Nakeeb — http://www.mans.edu.eg/en/ — through elnakeebayman@yahoo.com